CLINICAL TRIAL: NCT00785447
Title: Comparison of the Efficiency of Mouth-to-nose Breathing With Mouth-to-mouth Breathing in Non-paralyzed Adult Patients Under General Anesthesia
Brief Title: Comparison of the Efficiency of Mouth-to-nose Breathing With Mouth-to-mouth Breathing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Robert M. Kacmarek, Professor of Anesthesia, Director of Respiratory Care Services, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007-P-001680
Record Dates: First submitted 2008-10-30; First posted 2008-11-05 (Estimated); Last update posted 2012-04-25 (Estimated); Status verified 2012-04

CONDITIONS: Cardiopulmonary Resuscitation; Respiratory Physiology
Keywords: Cardiopulmonary Resuscitation; Respiratory Physiology; Mouth to mouth ventilation; Mouth to nose ventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other): Twenty healthy subjects between 18 to 59 years of age meeting ASA I-II criteria, undergoing elective surgery, requiring general anesthesia and being able to breathe through both their nose and mouth.
  Interventions: Other: Mouth-to-mouth or mouth-to-nose breathing

INTERVENTIONS:
Other: Mouth-to-mouth or mouth-to-nose breathing — Patients undergoing elective surgery under general anesthesia will be given mouth-to-mouth and mouth-to-nose breaths. The respiration process will be measured and recorded by the help of elastic bands put around the chest and abdomen. The efficiency of the breathing methods will be evaluated.

SUMMARY:
The purpose of this study is to find out the best way of providing artificial breathing during cardiopulmonary resuscitation (CPR). Current standard CPR involves giving mouth-to-mouth breathing to people requiring CPR. The rescuer pinches the person's nostrils closed and breathes into the mouth of the unconscious person with his or her own mouth.

Some CPR studies have shown that it might be easier and more effective to breathe air into a person's nose instead of the mouth. People receiving CPR often have blocked airways, so breathing into the mouth does not always work.

We think mouth-to-nose breathing may be more efficient and easier to do. In this case, the rescuer closes the person's mouth by pushing the jaw up and holding it still. Then the rescuer breathes into the unconscious person's nose by covering the nose entirely with his or her mouth. We are doing this study to try to find out which way works better.

We will perform both ways of breathing on people who are unconscious (asleep) before planned (non-emergency) surgery and compare their effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects between 18 to 59 years of age
* meeting ASA I-II criteria
* Undergoing elective surgery and requiring general anesthesia
* Being able to breathe through both the nose and the mouth while awake

Exclusion Criteria:

1. Patients with known infectious diseases, bacteria infections such as Neisseria meningitidis, upper respiratory tract infection (URI), bacterial pneumonia, etc. and patients with known HIV, HBV, HCV, or TB infection. Patients with broken oral mucosa or obvious sores.
2. Patients with immunosuppression from radiotherapy, chemotherapy, etc.
3. Patients with cardiovascular disease, respiratory disease, cerebral vascular disease and ASA class III or greater risk for anesthesia as defined by the American Society of Anesthesiologists.
4. Abnormal vital signs on the day of admission for surgery (HR, BP, room air oxygen saturation, EKG) that are not correctable with his or her routine medication or commonly used pre-operative medication.
5. Ischemic heart disease with chest pain or arrhythmias, patients with a pacemaker or AICD device and patients with heart failure.
6. Respiratory diseases, including subjects with COPD, asthma, pulmonary hypertension, restrictive lung disease, pleural effusion, tracheal stenosis and tracheal malacia, respiratory tract infection within the preceding week and those with previous pneumonectomy, lobectomy, tracheostomy, laryngectomy, tongue resection, and pharyngeal laryngeal plasity.
7. Unable to open mouth (<2.5 cm) or unable to breathe through mouth or nose.
8. Anticipated difficult airway: Mallampati score of III or greater, decreased neck movement, decreased mandibular movement, history of therapeutic radiation to the larynx or neck, prominent incisors. Subjects require or may require fiberoptic intubation
9. Important nasal septum deviation or other conditions impairing nasal breathing. The patient's nasal patency will be confirmed by inspiring with the mouth shut and open.
10. Gastric-esophageal reflex or a full stomach.
11. Obese with BMI greater than 35.
12. Neurological symptoms associated with neck extension, neurological deficit from previous stroke or spinal cord injury, recent stroke or TIA within 2 weeks.
13. Pregnant women and women less than one month post-partum. Ruling out pregnancy will be conducted by careful history and physical examination as done routinely prior to a surgery. If the history is believed to be unreliable, the patient will be excluded unless a pregnancy test is performed and the result of the test is negative.
14. Emergency cases, and subjects who have not adhered to the ASA NPO guidelines.
15. Prisoners.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2008-03; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Comparing CO2 elimination with mouth-to-nose versus mouth-to-mouth breathing in non-paralyzed adult patients under general anesthesia. | 1.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Yandong Jiang, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States